CLINICAL TRIAL: NCT02984436
Title: High-Sensitivity Cardiac Troponin T to OPtimize Chest Pain Risk Stratification
Acronym: STOP CP
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: STOP CP; OCR15652 (Other: University of Florida); 20162880 (Other: WIRB)
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Acute Coronary Syndrome; Chest Pain
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ED Patients with Acute Chest Pain: Emergency Department (ED) Patients with Acute Chest Pain will have blood samples collected for High sensitivity cardiac troponin T (hs-CTnT) analysis. Results from this analysis will be integrated into the HEART Score/Pathway. It will later be seen if integration of the hs-cTnT outperforms the use of HEART Score/Pathway alone.
  Interventions: Procedure: Blood Sample; Behavioral: HEART Score

INTERVENTIONS:
Procedure: Blood Sample — Blood samples will be collected from study participants for hs-cTnT analysis. Results of hs-cTnT will be used for research purposes only. Providers and participants will be blinded to results and participants will be treated by their healthcare providers per the standard of care.
  Other Names: Blood draw
Behavioral: HEART Score — The HEART Score is a prospectively studied scoring system to help emergency departments risk-stratify chest pain patients. Patients score on a scale of 0-10.
  Other Names: HEART Pathway

SUMMARY:
This is a prospective observational cohort study of ED patients with acute chest pain or other symptoms suggestive of ACS. Blood samples will be collected from study participants for High-Sensitivity Cardiac Troponin T (hs-cTnT) analysis. Results from hs-cTnT will be used for research purposes only.

Providers will be blinded to results and participants will be treated by their healthcare providers per the standard of care. Participants will have 30 and 90 day phone follow-ups to ascertain study outcomes.

DETAILED DESCRIPTION:
Approximately 8 million - 10 million patients complaining of chest pain present to an Emergency Department (ED) annually in the United States. To avoid missing the diagnosis of acute coronary syndrome (ACS), physicians use a liberal testing strategy. Thus, >50% of ED patients with acute chest pain are hospitalized for a comprehensive cardiac evaluation (serial cardiac biomarkers and stress testing or angiography). However, <10% of these patients are ultimately diagnosed with ACS, and this pervasive over-triage costs an estimated $10 billion - $13 billion annually. Current care patterns for acute chest pain fail to focus health system resources, such as hospitalization and stress testing, on patients most likely to benefit.

It has demonstrated that an accelerated diagnostic protocol (ADP), called the HEART Pathway, which utilizes a clinical decision aid (the HEART score) and serial Cardiac Troponin (cTn) measures are sensitive for ACS (>99%) and can substantially reduce hospitalizations, stress testing, and cost compared to usual care. The HEART Pathway uses contemporary serial cTn measurements at 0 and 3 hours to exclude index myocardial infarction (MI) and relies on clinical features (history, ECG, age, and risk factors) to identify patients likely to have downstream events. However, the HEART Pathway has limitations: a) It identifies only 20 - 40% of patients for early discharge and b) it was developed before high-sensitivity cTn assays became available. Able to detect MI earlier and with greater accuracy than contemporary assays, hs-cTn assays have the potential to be integrated into decision aids to improve chest pain risk stratification. In the near future, hs-cTn assays will replace contemporary assays in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 21 years at the time of enrollment in the ED
2. Chest discomfort or other symptoms consistent with possible ACS in which the treating physician plans to obtain an ECG and cTn for the patient's evaluation in the ED

Exclusion Criteria:

1. New ST-segment elevation consistent with myocardial infarction
2. Evidence of shock identified by the provider at the bedside and/or the PI
3. Terminal diagnosis with life expectancy less than 90 days
4. A non-cardiac medical, surgical, or psychiatric illness determined by the provider to require admission
5. Prior enrollment in the STOP CP study
6. Lack of capacity to provide consent and comply with study procedures
7. Inability to be reliably reached after the index visit for follow-up
8. Non-English speaking
9. Pregnant patients
10. Provider does not intend on obtaining serial cTn assays for evaluation of ACS
11. The first study draw (T0) will exceed 1 hour after the site-specific standard of care troponin draw
12. Unable or unwilling to authorize medical records release

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 21 years of age or older with possible Acute Coronary Syndrome (ACS) and associated chest pain.
Sampling Method: Non-Probability Sample
Enrollment: 1572 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
High Sensitivity Cardiac Troponin T using lithium heparin tubes | Baseline
  The research team will obtain two lithium heparin tubes at baseline, 1, 2, and 3 hours for sampling and preparation for shipping to the core laboratory in Maryland for hs-cTnT processing. Providers will be blinded to hs-cTnT results.
High Sensitivity Cardiac Troponin T using lithium heparin tubes | 1 hour after baseline
  The research team will obtain two lithium heparin tubes at baseline, 1, 2, and 3 hours for sampling and preparation for shipping to the core laboratory in Maryland for hs-cTnT processing. Providers will be blinded to hs-cTnT results.
High Sensitivity Cardiac Troponin T using lithium heparin tubes | 2 hours after baseline
  The research team will obtain two lithium heparin tubes at baseline, 1, 2, and 3 hours for sampling and preparation for shipping to the core laboratory in Maryland for hs-cTnT processing. Providers will be blinded to hs-cTnT results.
High Sensitivity Cardiac Troponin T using lithium heparin tubes | 3 hours after baseline
  The research team will obtain two lithium heparin tubes at baseline, 1, 2, and 3 hours for sampling and preparation for shipping to the core laboratory in Maryland for hs-cTnT processing. Providers will be blinded to hs-cTnT results.
High Sensitivity Cardiac Troponin T using EDTA tubes | Baseline
  The research team will obtain one EDTA tube at baseline, 1, 2, and 3 hours for sampling and preparation for shipping to the core laboratory in Maryland for hs-cTnT processing. Providers will be blinded to hs-cTnT results.
High Sensitivity Cardiac Troponin T using EDTA tubes | 1 hour after baseline
  The research team will obtain one EDTA tube at baseline, 1, 2, and 3 hours for sampling and preparation for shipping to the core laboratory in Maryland for hs-cTnT processing. Providers will be blinded to hs-cTnT results.
High Sensitivity Cardiac Troponin T using EDTA tubes | 2 hours after baseline
  The research team will obtain one EDTA tube at baseline, 1, 2, and 3 hours for sampling and preparation for shipping to the core laboratory in Maryland for hs-cTnT processing. Providers will be blinded to hs-cTnT results.
High Sensitivity Cardiac Troponin T using EDTA tubes | 3 hours after baseline
  The research team will obtain one EDTA tube at baseline, 1, 2, and 3 hours for sampling and preparation for shipping to the core laboratory in Maryland for hs-cTnT processing. Providers will be blinded to hs-cTnT results.
Cardiac Troponin T (cTn) | Baseline
  Site-specific cTn will be measured at baseline
Cardiac Troponin T (cTn) | 3 hours
  Site-specific cTn will be measured at 3 hours unless baseline site-specific cTn tests positive
Occurrence of major adverse cardiac events (MACE) | 30 days
Occurrence of major adverse cardiac events (MACE) | 90 days

SECONDARY OUTCOMES:
HEART Score Calculation | Change from Baseline, 1, 2, 3 hours. 30 days and 90 days post discharge
  By assigning zero, one, or two points - towards an atypical patient history, ECG anomalies, the patient's age, any risk factors present, and elevated Troponin - patients score on a scale of 0-10. 0-3 = Low-risk, 4 or greater = High-risk
Incidence and Intensity of Adverse Events | Change from Baseline, 1, 2, 3 hours. 30 days and 90 days post discharge
  Number of Participants with treatment related Adverse Events as Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Brandon R Allen, MD, Principal Investigator — University of Florida
Locations (6):
- United States (6):
  - UC Davis, Sacramento, California
  - University of Florida, Gainesville, Florida
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashburn NP, Snavely AC, Supples MW, Millard MJ, Allen BR, Christenson RH, Madsen T, Mumma BE, Hashemian T, Wilkerson RG, Mahler SA. Performance of the High-STEACS Early Rule Out Pathway Using hs-cTnT at 30 Days in a Multisite US Cohort. Circ Cardiovasc Qual Outcomes. 2025 Feb;18(2):e011084. doi: 10.1161/CIRCOUTCOMES.124.011084. Epub 2025 Jan 9. PMID 39781769
- [Derived] Supples MW, Dameron AG, Powell S, Snavely AC, Ashburn NP, Allen BR, Christenson RH, Wilkerson RG, Mumma BE, Madsen TE, Mahler SA. The HET (history, electrocardiogram, and troponin) score has low efficacy and negative predictive value in a multisite U.S. cohort study. Am J Emerg Med. 2025 Mar;89:151-158. doi: 10.1016/j.ajem.2024.12.012. Epub 2024 Dec 15. PMID 39729682
- [Derived] Millard MJ, Ashburn NP, Snavely AC, Hashemian T, Supples M, Allen B, Christenson R, Madsen T, McCord J, Mumma B, Stopyra J, Wilkerson RG, Mahler SA. European Society of Cardiology 0/1-hour algorithm (high-sensitivity cardiac troponin T) performance across distinct age groups. Heart. 2024 May 23;110(12):838-845. doi: 10.1136/heartjnl-2023-323621. PMID 38471727
- [Derived] Ashburn NP, Snavely AC, Allen BR, Christenson RH, Madsen T, McCord JK, Mumma BE, Hashemian T, Stopyra JP, Wilkerson RG, Mahler SA. Performance of the European Society of Cardiology 0/1-hour algorithm with high-sensitivity cardiac troponin T at 90 days among patients with known coronary artery disease. Am J Emerg Med. 2024 May;79:111-115. doi: 10.1016/j.ajem.2024.02.029. Epub 2024 Feb 23. PMID 38417221
- [Derived] Supples MW, Snavely AC, O'Neill JC, Ashburn NP, Allen BR, Christenson RH, Nowak R, Wilkerson RG, Mumma BE, Madsen T, Stopyra JP, Mahler SA. Sex and race differences in the performance of the European Society of Cardiology 0/1-h algorithm with high-sensitivity troponin T. Clin Cardiol. 2024 Feb;47(2):e24199. doi: 10.1002/clc.24199. Epub 2023 Dec 13. PMID 38088463
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Aldous SJ, Allen BR, Apple FS, Babel H, Christenson RH, Cullen L, Di Carluccio E, Doudesis D, Ekelund U, Giannitsis E, Greenslade J, Inoue K, Jernberg T, Kavsak P, Keller T, Lee KK, Lindahl B, Lorenz T, Mahler SA, Mills NL, Mokhtari A, Parsonage W, Pickering JW, Pemberton CJ, Reich C, Richards AM, Sandoval Y, Than MP, Toprak B, Troughton RW, Worster A, Zeller T, Ziegler A, Blankenberg S; ARTEMIS study group. Personalized diagnosis in suspected myocardial infarction. Clin Res Cardiol. 2023 Sep;112(9):1288-1301. doi: 10.1007/s00392-023-02206-3. Epub 2023 May 2. PMID 37131096
- [Derived] Allen BR, Christenson RH, Cohen SA, Nowak R, Wilkerson RG, Mumma B, Madsen T, McCord J, Huis In't Veld M, Massoomi M, Stopyra JP, Montero C, Weaver MT, Yang K, Mahler SA. Diagnostic Performance of High-Sensitivity Cardiac Troponin T Strategies and Clinical Variables in a Multisite US Cohort. Circulation. 2021 Apr 27;143(17):1659-1672. doi: 10.1161/CIRCULATIONAHA.120.049298. Epub 2021 Jan 21. PMID 33474976